CLINICAL TRIAL: NCT07105111
Title: A Phase 4, Open-Label Study to Evaluate the Efficacy of Valbenazine on Clinician- and Patient-Reported Outcomes in Patients With Tardive Dyskinesia (TD) Who Remain Symptomatic While on Deutetrabenazine or After Discontinuing Prior TD Treatment With a Vesicular Monoamine Transporter 2 (VMAT2) Inhibitor
Brief Title: A Study to Evaluate the Effectiveness of Valbenazine in Adult Participants With Tardive Dyskinesia (TD) Who Remain Symptomatic While Receiving or After Stopping a Vesicular Monoamine Transporter 2 (VMAT2) Inhibitor
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBI-98854-TD4027
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder; Major Depressive Disorder; Tardive Dyskinesia
Keywords: Valbenazine
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder; Depressive Disorder, Major; Tardive Dyskinesia | interventions — valbenazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Valbenazine (Experimental): Valbenazine administered once daily for 24 weeks.
  Interventions: Drug: Valbenazine

INTERVENTIONS:
Drug: Valbenazine — Valbenazine capsules for oral administration.
  Other Names: NBI-98854

SUMMARY:
This study will evaluate the efficacy of valbenazine on clinician- and patient-reported outcomes in participants with TD while receiving or after stopping a VMAT2 inhibitor.

ELIGIBILITY:
Key Inclusion Criteria:

* 18 years of age or older
* Diagnosed with one of the following at least 3 months prior to screening: schizophrenia or schizoaffective disorder, bipolar disorder, or major depressive disorder
* Diagnosed with at least mild neuroleptic-induced TD for at least 3 months prior to screening

Key Exclusion Criteria:

* Have comorbid Parkinsonism or abnormal involuntary movement(s) that is more prominent than TD
* Diagnosis of moderate or severe substance use disorder in the last 6 months
* History of long QT syndrome, cardiac arrythmia, or severe hepatic impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-29 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Abnormal Involuntary Movement Scale (AIMS) Dyskinesia Total Score (AIMS 1-7) at Week 24 | Baseline, Week 24

SECONDARY OUTCOMES:
Change from Baseline in the Clinical Global Impression of Severity - Tardive Dyskinesia (CGI-TD-S) Score at Week 24 | Baseline, Week 24
Change from Baseline in the Tardive Dyskinesia Impact Scale (TDIS) at Week 24 | Baseline, Week 24
Change from Baseline in the EuroQol-Visual Analogue Scale (EQ-VAS) at Week 24 | Baseline, Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Lead, Study Director — Neurocrine Biosciences
Locations (8):
- United States (8):
  - Neurocrine Clinical Site, Bryant, Arkansas
  - Neurocrine Clinical Site, Fountain Valley, California
  - Neurocrine Clinical Site, Orange, California
  - Neurocrine Clinical Site, Bonita Springs, Florida
  - Neurocrine Clinical Site, Hialeah, Florida
  - Neurocrine Clinical Site, Miami, Florida
  - Neurocrine Clinical Site, Tampa, Florida
  - Neurocrine Clinical Site, Marietta, Georgia